CLINICAL TRIAL: NCT03386903
Title: Acupuncture Regulates Emotion-cognitive Network of Chronic Insomnia Patients : A DTI-fMRI Study
Brief Title: Acupuncture Regulates Default Mode Network of Chronic Insomnia Disorder Patients : A fMRI Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Ping Zhou, Principal Investigator, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016BL-033-01
Record Dates: First submitted 2017-08-09; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ture acupuncture group (Experimental): After recruiting, patients are assigned to the ture acupuncture group by randomization,and then receive ture acupuncture treatment. patients are scanned by MRI at the baseline and 3 month post-treatment respectively.
  Interventions: Device: Ture acupuncture
- Sham acupuncture group (Placebo Comparator): After recruiting, patients are assigned to the sham acupuncture group by randomization,and then receive sham acupuncture stimulation. patients are scanned by MRI at the baseline and 3 month post-treatment respectively.
  Interventions: Device: Sham acupuncture
- Healthy group (No Intervention): Healthy subjects without intervention except scanned brain image by MRI at the baseline.

INTERVENTIONS:
Device: Ture acupuncture — Patients receive true acupuncture treatment by Zhoushi coordinated points at the "Bai-hui" (DU20), "Shen-ting" (DU24), bilateral "Ben-shen" (BG13), "Shen-men" (HT7), "San-yin-jiao" (SP6) with "Deqi" sensation. The needles are retained for 20 minutes in every course, three times per week and last for 3 months.
  Other Names: Experimental
  Arms: Ture acupuncture group
Device: Sham acupuncture — Patients receive sham acupuncture stimulation by non-acupoint points (superficial insertion, 0.2 cun, No needle sensation (de qi) is elicited) at the bilateral mid-point between Shuaigu(GB8) and Touwei(ST8), Touwei(ST8) and Yangbai(GB14), front tibia, the junction of biceps and triceps.
  Other Names: Placebo Comparator
  Arms: Sham acupuncture group

SUMMARY:
The purpose of the study is to investigate the underlying central nervous mechanisms of acupuncture treatment in chronic insomnia patients, from observation changes of gray matter and functional connectivity in the default mode network and the salience network by functional magnetic resonance imaging, and combine with clinical efficacy assessment to analyze the association between the results of imaging and behavioristic.

DETAILED DESCRIPTION:
Chronic insomnia which can cause daytime function impairments like abnormal emotion and hypomnesis is important risk factors for developing cardiovascular disease, neurological disorders or mental disorders. Acupuncture is a widely recognized therapy to treat chronic insomnia in clinical practice. Previous researches presented that sleep-wake dysfunction of patients with chronic insomnia have strong correlation with abnormal of the default mode network and salience network. The project present acupuncture may improve sleep quality by adjusting the abnormal default mode network and the salience network in patients with chronic insomnia.

The investigators are assigned the ninety eligible participants in three groups: thirty chronic insomnia patients by true acupuncture treatment (Zhoushi coordinated points), thirty chronic insomnia patients by sham acupuncture stimulation (non-acupoint points) and thirty healthy subjects, Treatment will be given 3 times per week for 3 months. Additionally, two methods include functional magnetic resonance imaging (fMRI) and clinical scales evaluation as the outcome measures to evaluate the effectiveness and security of acupuncture. Outcomes will be evaluated at baseline and 3 month post-treatment.

The aim of this project is to investigate effect of acupuncture treatment on gray matter and functional connectivity of the default network and the salience network in chronic insomnia patients, and to analyze the association between sleep quality, emotion, day function with imaging results. The central nervous mechanisms underlying acupuncture treatment are discussed by this finding which may provide scientific basis for acupuncture treatment in chronic insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia group: Patients must meet DSM V criteria for chronic insomnia. PSQI>7 、ISI>7、 SAS<50、 SDS<50.
* control group: no self-reported sleep problems in the last 1 months. PSQI≤5 、SAS<50、 SDS<50，MMSE≥27.
* 30-60 years old.
* Male or female.
* Dextromanuality.
* Having given written informed consent to participate in the research project.

Exclusion Criteria:

* History of cardiovascular and respiratory diseases.
* Other diagnoses of the nerve or mental disorders.
* Other sleep disorders.
* The long history of smoking, drinking and abusing drugs, or taking psychotropic drugs in last month, and treatment in other clinical trials at the same time.
* The body carrying pacemakers, defibrillators, implantable vascular clamp, implantable electric or magnetic device, mechanical heart valve, artificial cochlear, el., fMRI taboo and the claustrophobic.
* MRI scans have been used to identify patients with a definite organic lesion or severe head anatomical asymmetry
* Pregnancy, lactation and peri menopausal women.
* An allergy history of syncope, alcohol, and metal needle.
* The body Mass Index>32 or <19.8.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-02-28 (Estimated); Primary Completion 2018-12-28 (Estimated); Study Completion 2019-06-28 (Estimated)

PRIMARY OUTCOMES:
Sleep quality obtained by questionnaire:Pittsburgh Sleep Quality Index | baseline,12 weeks
  Change in Pittsburgh sleep quality index scores at the baseline and the end of 12 weeks stimulation with acupuncture.Minimum Score = 0 (good sleep); Maximum Score = 30 (disrupted sleep)

SECONDARY OUTCOMES:
Brain gray matter | baseline,12 weeks
  The changes of gray matter volume in default network before and after treatment
Total sleep time obtained by questionnaire:Pittsburgh Sleep Quality Index | baseline,12 weeks
Sleep efficiency obtained by questionnaire:Pittsburgh Sleep Quality Index | baseline,12 weeks
Sleep latency obtained by questionnaire:Pittsburgh Sleep Quality Index | baseline,12 weeks
Wake after sleep onset obtained by questionnaire:Pittsburgh Sleep Quality Index | baseline,12 weeks
Sleep problem obtained by questionnaire:Insomnia Severity Index | baseline,12 weeks
Emotional state of anxiety obtained by questionnaire:Self-Rating Anxiety Scale | baseline,12 weeks
Emotional state of depression obtained by questionnaire:Self-Rating Depression Scale | baseline,12 weeks
Daytime function obtained by questionnaire:Epworth Sleepiness Score | baseline,12 weeks
Daytime function obtained by questionnaire:Flinders Fatigue Scale | baseline,12 weeks
resting-state functional magnetic resonance imaging | baseline,12 weeks
  Resting state intrinsic connectivity within the default network by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Liu cun zhi, M.D, Study Director — Beijing Hospital of Traditional Chinese Medicine
Locations (1):
- Beijing Hostipal of Traditional Chinese Medicine affiliated to Capital medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided